CLINICAL TRIAL: NCT03570021
Title: ESTIMation of the ABiLity of Prophylactic Central Compartment Neck Dissection to Modify Outcomes in Low-risk Differentiated Thyroid Cancer
Acronym: ESTIMABL3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A01779-44; 2017/2581 (Other: CSET number)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Neck Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): total thyroidectomy with bilateral prophylactic central compartment (level VI) neck dissection as defined by the American Thyroid Association [American Thyroid Association Surgery Working Group, Thyroid 2009]. This is a standard treatment recognized by the French Society of Otolaryngology Head and Neck Surgery [French Society of Otolaryngology Head and Neck Sugery].
  Interventions: Procedure: total thyroidectomy with bilateral prophylactic central compartment (level VI) neck dissection
- Group 2 (Experimental): total thyroidectomy alone without neck dissection. This is recognized as a standard treatment by the Francophone Association of Endocrine Surgery
  Interventions: Procedure: total thyroidectomy alone without neck dissection

INTERVENTIONS:
Procedure: total thyroidectomy with bilateral prophylactic central compartment (level VI) neck dissection — total thyroidectomy with bilateral prophylactic central compartment (level VI) neck dissection as defined by the American Thyroid Association [American Thyroid Association Surgery Working Group, Thyroid 2009]. This is a standard treatment recognized by the French Society of Otolaryngology Head and Neck Surgery [French Society of Otolaryngology Head and Neck Sugery].
  - The number of lymph nodes resected, the number of metastatic nodes, their size and the presence or absence of extranodal spread will be recorded. Due to the large natural variability of the number of lymph nodes retrieved in a prophylactic neck dissection [Hartl DM, Ann Surg 2012], no patient will be excluded on the basis of number of lymph nodes. Furthermore, the participating surgeons routinely perform complete central neck dissections, and were chosen to participate in this study due to a homogenous technique among these surgeons [Hartl DM, World J Surg 2012].
  Arms: Group 1
Procedure: total thyroidectomy alone without neck dissection — This is recognized as a standard treatment by the Francophone Association of Endocrine Surgery
  Arms: Group 2

SUMMARY:
Prospective randomized open phase III non-inferiority trial in cT1bT2N0 papillary thyroid carcinoma comparing: total thyroidectomy alone (experimental group) versus total thyroidectomy + Prophylactic Neck Dissection PND (reference group).

Pre-registered patients will be randomized before surgery for tumors with class-6 cytology (Bethesda) or in the operating room after confirmation of malignancy by frozen section analysis for tumors with class-5 cytology.

ELIGIBILITY:
Inclusion Criteria:

1. Thyroid nodule measuring 11-40 mm on ultrasound (cT1bT2)

   * AND with fine-needle aspiration biopsy (FNAB) cytology in favor of "papillary thyroid carcinoma" (Type 6 according to the Bethesda classification (Appendix 2)
   * OR with FNAB cytology "suspicious for malignancy" (Type 5 according to the Bethesda classification). In this latter case, randomization will be performed if confirmation of papillary carcinoma on intraoperative frozen section analysis
2. cN0: absence of lymph nodes suspicious for malignancy on preoperative ultrasound performed by the center's designated radiologist according to a standardized report
3. Absence of a medical contra indication to performing a total thyroidectomy with or without bilateral prophylactic neck dissection of the central compartment
4. Women of childbearing potential should have a negative pregnancy test (serum or urine) before any radioiodine administration. Sexually active patients must agree to use an effective method of contraception or to abstain from sexual activity during the study and for at least 6 months after last dose of radioiodine.
5. Patient affiliated to a social security regimen or beneficiary of such regimen
6. Patients age ≥ 18 years old, french-speaking
7. Patients should understand, sign and date the written informed consent form prior to any protocol specific procedures. Patients should be able and willing to comply with study visits.

Exclusion Criteria:

1. Tumors > 40 mm (cT3) or ≤ 10 mm
2. Tumors with extrathyroidal extension suspected or obvious on the pre-operative work-up or intra-operatively (cT3T4)
3. Metastatic neck lymph nodes or suspicious neck nodes on preoperative ultrasound (cN1); for suspicious nodes, FNAB cytology and thyroglobulin assay on the needle washout fluid will be performed
4. Metastatic neck lymph nodes found during the thyroidectomy and confirmed with intra-operative frozen section analysis
5. Medullary thyroid carcinoma on FNAB cytology and/or with basal serum calcitonin >50 pg/ml
6. Preoperative or intra-operative suspicion of non-papillary thyroid carcinoma or aggressive histopathological subtype or poorly differentiated carcinoma
7. Distant metastases (M1) apparent pre-operatively (found due to symptoms or fortuitously; no specific pre-operative work-up will be performed, however, in accordance with current clinical practice)
8. Recurrent nerve paralysis visualized on systematic pre-operative laryngoscopy and/or abnormal preoperative serum calcium
9. Pregnant or breast feeding women
10. Participation in another therapeutic clinical trial within one year from study entry
11. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients in complete remission | 1 year after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hartl D, Godbert Y, Carrat X, Bardet S, Lasne-Cardon A, Vera P, Ilies E, Zerdoud S, Sarini J, Zalzali M, La Manna L, Schneegans O, Kelly A, Kauffmann P, Rodien P, Brunaud L, Grunenwald S, Housseau E, Laghouati S, Bouvet N, Lecerf E, Hadoux J, Lamartina L, Schlumberger M, Borget I. ESTIMation of the ABiLity of prophylactic central compartment neck dissection to modify outcomes in low-risk differentiated thyroid cancer: a prospective randomized trial. Trials. 2023 Apr 28;24(1):298. doi: 10.1186/s13063-023-07294-0. PMID 37118818